CLINICAL TRIAL: NCT01882101
Title: Comparison of Posterior Tibial Nerve Stimulation and Biofeedback for Fecal Incontinence: Prospective Randomized Controlled Trial
Brief Title: Comparison of PTNS and Biofeedback for Fecal Incontinence
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Too small included patients and, not enough cost for PTNS and biofeedback.
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); National Cancer Center, Korea (Other Government); Seoul National University Boramae Hospital (Other); Hallym University Medical Center (Other); Daehang Hospital (Other)
Responsible Party: Principal Investigator, Sung-Bum Kang, Principal Investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTNS trial
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; posterior tibial nerve stimulation; biofeedback; quality of life
MeSH Terms: conditions — Fecal Incontinence | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior tibial nerve stimulation (Experimental)
  Interventions: Procedure: Posterior tibial nerve stimulation
- Biofeedback (Experimental)
  Interventions: Procedure: Biofeedback

INTERVENTIONS:
Procedure: Posterior tibial nerve stimulation — 34G needle is introduced percutaneously three finger-breadths superior to the medial malleolus and an electrode is attached to the ipsilateral foot. Electrical stimulation is applied monitoring motor and sensory response. The treatment lasts for 30 minutes, and will be repeated twice a week for 6 weeks.
  Other Names: PTNS
  Arms: Posterior tibial nerve stimulation
Procedure: Biofeedback — Electrodes are attached to the lower abdomen and acryl plug is inserted into the anal canal. The patients perform pelvic muscle exercise watching EMG activity of themselves. The treatment lasts over 30 minutes, and will be repeated twice a week for 6 weeks.
  Other Names: Pelvic floor muscle exercise
  Arms: Biofeedback

SUMMARY:
Until recently, there is no definite treatment for fecal incontinence that is proven to be effective with low morbidity. The efficacy of biofeedback therapy for incontinence has not been proven on the randomized controlled trials. Sacral nerve stimulation is too expensive although some prospective studies showed the therapeutic potential. Recently, posterior tibial nerve stimulation has been reported to be effective with lower cost in comparison with sacral nerve stimulation. This study is designed to show the efficacy of posterior tibial nerve stimulation compared with biofeedback therapy for fecal incontinence.

DETAILED DESCRIPTION:
This prospective randomized controlled trial is designed to compare the efficacy of biofeedback and posterior tibial nerve stimulation for fecal incontinence. Primary endpoint is weekly episodes of fecal incontinence at 1 week after each treatment. Sample size was calculated as 50 patients. Outcomes include weekly episodes and severity of fecal incontinence, quality of life and anal function. Outcomes will be assessed using bowel diary, FISI questionnaire, FIQL questionnaire and anorectal manometry at 1,8,16 and 24 weeks after each treatment for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient with 2 or more weekly episodes of fecal incontinence
* Patient who understands and accepts to sign the informed consent form

Exclusion Criteria:

* Patient with gas incontinence only
* Major injury in anal sphincter
* Anorectal operation history within 24 months
* Previous spinal injury, tumor or surgery
* Presence of neurological disease
* Peripheral vascular disease
* Severe comorbidity
* Psychiatric disorder
* Legally prohibited for clinical trial
* Pregnancy or breast feeding
* Previous disease or disability expected to influence the assessment of postoperative quality of life

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Weekly episodes of fecal incontinence | 1 week
  Measured by bowel diary at pre-treatment(baseline) and post-treatment(1 week)

SECONDARY OUTCOMES:
Weekly episodes of fecal incontinence | 6 months
  Measured by bowel diary at post-treatment(2, 4, 6 months)
Severity of fecal incontinence | 6 months
  Measured by FISI questionnaire at pre-treatment(baseline) and post-treatment(1 week, 2, 4, 6 months)
Quality of life associated with fecal incontinence | 6 months
  Measured by FIQL questionnaire at pre-treatment(baseline) and post-treatment(1 week, 2, 4, 6 months)
Anal function | 6 months
  Measured by manometry at pre-treatment(baseline) and post-treatment(1 week, 2, 4, 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bum Kang, Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (6):
- South Korea (6):
  - Hallym University College of Medicine, Anyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Daehang Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul